CLINICAL TRIAL: NCT02103894
Title: Evaluation of [18F]MNI-777 PET as a Marker of Tau Pathology in Subjects With Clinically Diagnosed Tauopathies in Comparison to Healthy Subjects
Brief Title: Evaluation of [18F]MNI-777 PET as a Marker of Tau Pathology in Subjects With Tauopathies Compared to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Molecular NeuroImaging (Other)
Collaborators: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Principal Investigator, Danna Jennings, Principal Investigator, Molecular NeuroImaging
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: MNI-777
Record Dates: First submitted 2014-02-12; First posted 2014-04-04 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Alzheimer's Disease (AD); Parkinson's Disease (PD); Chronic Traumatic Encephalopathy (CTE); Progressive Supranuclear Palsy (PSP); Frontal Temporal Dementia (FTD); Pick's Disease; Tauopathies
Keywords: Alzheimer's disease (AD); Parkinson's disease (PD); Progressive supranuclear palsy (PSP); Chronic traumatic encephalopathy (CTE); Frontal temporal dementia (FTD); Pick's disease; tauopathies
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease; Chronic Traumatic Encephalopathy; Supranuclear Palsy, Progressive; Pick Disease of the Brain; Tauopathies | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole; florbetapir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [18F]T807 ([18F]MNI-777) (Experimental): At the [18F]MNI-777 PET imaging visit, subjects will be injected with no more than 10 mCi (370 MBq) of [18F]MNI-777).
  Interventions: Drug: [18F]T807 ([18F]MNI-777)

INTERVENTIONS:
Drug: [18F]T807 ([18F]MNI-777) — All enrolled subjects will undergo an [18F]MNI-777 PET imaging visit. For individuals with AD or CTE, [18F]florbetapir imaging may also be performed to serve as a means of correlating disease severity by evaluating the relationship of β-amyloid uptake (measured by [18F]florbetapir imaging) and tau protein uptake (measured by [18F]MNI-777 PET imaging). For individuals with Parkinsonian symptoms, [123I]β-CIT SPECT imaging may be performed to evaluate for a reduction in dopamine transporter uptake.
  Other Names: [18F]T807; [18F]florbetapir; Amyvid; [123I]β-CIT

SUMMARY:
The goal of this study is to assess [18F]MNI-777 PET imaging as a tool to detect tau pathology in the brain of individuals who carry a clinical diagnosis of a tauopathy, including: Alzheimer's Disease (AD),Parkinson's disease (PD) Progressive Supranuclear Palsy (PSP), chronic traumatic encephalopathy (CTE) and Frontal Temporal Dementia (FTD) and age- and gender-matched healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

For all subjects:

* Written informed consent or assent is obtained.
* Willing and able to cooperate with study procedures.
* For females, non-child bearing potential or negative urine pregnancy test on day of [18F]MNI-777 injection.

Alzheimer Disease subjects:

* The participant is 50 years or older.
* Participants have a clinical diagnosis of Alzheimer's disease based on National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria (McKann, 1984)
* Modified Hachinski Ischemia Scale score of ≤ 4.

Parkinson's Disease subjects:

* The participant is 30 years or older.
* Participants have a clinical diagnosis of PD based on the UK Brain Bank Criteria (Hughes, et al., 1982).
* The duration of diagnosis of PD is <20 years prior to the imaging visit
* PD subjects must be on stable doses of medications for a period of at least 30 days prior to the imaging visit.
* Treatment with dopamine replacement therapies or other symptomatic therapies for PD is permitted; however, subjects must be on a stable dose of medications 30 days prior to the imaging visit.

Progressive Supranuclear Palsy subjects:

* The participant is 30 years or older.
* Participants have a clinical diagnosis of PSP based on National Institute of Neurological Disorders and Stroke/ (NINDS) and the Society for PSP (SPSP) criteria (Litvan, et al. 1996).

Chronic Traumatic Encephalopathy subjects:

* The participant is 18 years or older.
* Subjects with a diagnosis of probable CTE based on a prior history of repetitive brain trauma and at least one concussion, and a current mood disorder (depression, apathy, irritability, suicidal ideation), cognitive symptoms (memory loss, impaired executive function) or behavioral symptoms (disinhibition, aggression and increased violence) (Jordan, 2013).

Frontal Temporal Dementia/Pick's disease subjects:

* The participant is 50 years or older.
* Participants have a clinical diagnosis of FTD based on consensus for clinical diagnosis of frontotemporal dementia (Neary, et al., 1998)

Healthy Control subjects:

* The participant is 18 - 85 years old.
* Negative history of neurological or psychiatric illness based on evaluation by a research physician.
* MMSE score must be 29 or above.

Exclusion Criteria:

All subjects will be excluded from participation for the following reasons:

* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness.
* The subject has any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including gastrointestinal surgery).
* The subject has evidence of a structural lesion on MRI that may interfere with interpretation of PET imaging.
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* The subject has participated in another clinical study within the previous 30 days.
* Pregnancy or women who are nursing or breastfeeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-02; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Brain uptake of [18F]T807 ([18F]MNI-777) | 2 years
  To quantitatively assess the brain uptake of [18F]MNI-777 ([18F]T807), an imaging biomarker for tau pathology in brain, using positron emission tomography (PET) in individuals with clinically diagnosed tauopathies including: Alzheimer's disease (AD), Parkinson's disease (PD), progressive supranuclear palsy (PSP), chronic traumatic encephalopathy (CTE) and frontal temporal dementia/Pick's disease (FTD) and healthy controls (HC).

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Molecular NeuroImaging, LLC, New Haven, Connecticut, United States

REFERENCES:
- [Background] Jordan BD. The clinical spectrum of sport-related traumatic brain injury. Nat Rev Neurol. 2013 Apr;9(4):222-30. doi: 10.1038/nrneurol.2013.33. Epub 2013 Mar 12. PMID 23478462
- [Background] McKhann G, Drachman D, Folstein M, Katzman R, Price D, Stadlan EM. Clinical diagnosis of Alzheimer's disease: report of the NINCDS-ADRDA Work Group under the auspices of Department of Health and Human Services Task Force on Alzheimer's Disease. Neurology. 1984 Jul;34(7):939-44. doi: 10.1212/wnl.34.7.939. PMID 6610841
- [Background] Litvan I, Agid Y, Calne D, Campbell G, Dubois B, Duvoisin RC, Goetz CG, Golbe LI, Grafman J, Growdon JH, Hallett M, Jankovic J, Quinn NP, Tolosa E, Zee DS. Clinical research criteria for the diagnosis of progressive supranuclear palsy (Steele-Richardson-Olszewski syndrome): report of the NINDS-SPSP international workshop. Neurology. 1996 Jul;47(1):1-9. doi: 10.1212/wnl.47.1.1. PMID 8710059
- See also: Molecular NeuroImaging — http://www.mnimaging.com
- See also: Institute for Neurodegenerative Disorders — http://www.indd.org